CLINICAL TRIAL: NCT02187614
Title: A Double Blind, Multi-arm Randomized Control Trial, for Efficacy of Intramuscular Diclofenac Versus Intravenous Morphine Versus Intravenous Paracetamol, in Renal Colic Emergency Department Pain Management
Brief Title: Efficacy Study of Different Analgesic Options in Kidney Stone Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. SAMEER PATHAN, Research Fellow and Specialist, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB Number: 14-00059; Hamad Medical Corporation-MRC (Other Grant/Funding Number: IRGC-01-NI-045)
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Renal Colic; Urinary Calculi
Keywords: Acute Renal colic; Acute Ureteric Colic; Renal or Ureteral Calculi; Urolithiasis; Kidney or Ureteral stones
MeSH Terms: conditions — Renal Colic; Urinary Calculi; Ureteral Calculi; Urolithiasis | interventions — Diclofenac; Morphine; Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diclofenac and Placebos (Experimental): Participants in this group will receive a Diclofenac 75 mg intramuscular injection, and two placebo saline solutions intravenously.
  Interventions: Drug: Diclofenac; Drug: Placebos
- Morphine and Placebos (Active Comparator): Participants in this group will receive Morphine 0.1 mg/kg intravenously, along with an additional intravenous placebo and an intramuscular placebo injection.
  Interventions: Drug: Morphine; Drug: Placebos
- Paracetamol and Placebos (Active Comparator): participants in this group will receive intravenous Paracetamol 1 gm solution, along with an additional intravenous placebo and an intramuscular placebo injection.
  Interventions: Drug: Paracetamol; Drug: Placebos

INTERVENTIONS:
Drug: Diclofenac
  Other Names: Voltaren; Diclofen; Diclorex
  Arms: Diclofenac and Placebos
Drug: Morphine
  Other Names: Morphine sulphate
  Arms: Morphine and Placebos
Drug: Paracetamol
  Other Names: Perfalgan; Acetaminophen
  Arms: Paracetamol and Placebos
Drug: Placebos
  Other Names: saline solution

SUMMARY:
Abdominal pain is one of the most common presentations to an emergency department (ED). Among patients presenting with abdominal pain, a common diagnosis in the Middle East is renal colic (urolithiasis or Kidney stones). As the patients with renal colic writhe around in agonizing pain, the first priority in an ED from a patient's perspective is fast and safe analgesia and to be pain free as early as possible. There are variations in physician preference to choose initial analgesic drug for managing such pain. Commonly used drugs are:

* Opioids such as Morphine or Fentanyl
* Non steroidal drugs such as Diclofenac, Ketorolac or Brufen
* and Paracetamol intravenous injection.

A robust evidence in comparison of diclofenac versus morphine and paracetamol is lacking. This study is design to obtain data on efficacy of these three drugs within 30 minutes in a non inferiority trail.

DETAILED DESCRIPTION:
This will be a double blind RCT, where participants will be enrolled consecutively after meeting eligibility criteria and obtaining a written informed consent. They will be assign to one of the three study arms by computer generated randomization process. The study packets will be prepared by a dedicated nurse or pharmacist who will not a part of investigating team. Each Patients will receive one analgesic drug (active drug) and two placebos. Drugs will be given as one intramuscular injection and two intravenous solutions.

Pain score will be recorded using NRS at 0, 30, 60, and 90 minutes. Data will be collected on standard Data collection form. Each participant will receive analgesia from study packet which contains, one active drug and two placebos to be administer as one intramuscular and two intravenous solutions. At any given time every patient will receive one analgesia from either Diclofenac, Paracetamol or Morphine. If patient pain does not respond to initial treatments, at 30 minutes a rescue analgesia in form of morphine will be administered till patient is pain free or NRS<=2 or adverse event to morphine.

Based on the results of previous studies (1-3), proportion of patients achieving more than 50% pain reduction, is between 65-75% for diclofenac, morphine and paracetamol when compared with other drugs. In each group, 437 patients are required to detect a difference of 10% in primary outcome, in a superiority trial with power (1-beta) of 90% and significance level (alpha) of 5% in this study. Considering 15% extra, total sample size required in this superiority trial will be 1507 patients in total.

Data will be collected on a standard data recording form and it will be converted to electronic excel sheet hiding patient identifiable details. Continuous variables will be presented as mean with standard deviation (SD). Categorical variables will be calculated as proportions and presented with 95% Confidence interval (CI). Statistical analyses will be undertaken using Stata 12.0 (College Station, Texas).

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years and < 65 years
* Acute onset, one side flank or loin pain, with or without radiation to groin or genital areas.
* Pain intensity on NRS more than or equal to 4. (Moderate to Severe Pain)
* Diagnosis confirmed by non contrast CT KUB within the ED visit.

Exclusion Criteria:

* Traumatic flank pain
* Pregnancy
* Known renal failure or impairment
* Known allergy to morphine, diclofenac or paracetamol
* Bronchial asthma
* Previously enrolled in the study.
* Use of any analgesia in last 6 hour.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1645 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving a reduction of >50% on Numerical Rating Scale (NRS-11) from the initial NRS recorded at the end of 30 minutes in each study arm. | at 30 minutes after analgesia

SECONDARY OUTCOMES:
reduction in mean NRS | at 30, 60 and 90 minutes after analgesia

OTHER OUTCOMES:
adverse event rate | Within 14 days of ED visit
total analgesia requirement to get pain score (NRS) less than or equal to 2. | by 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Sameer A. Pathan, MBBS, MCEM, Principal Investigator — Hamad Medical Corporation; Prof. Peter A Cameron, MD,FACEM, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Emergency Department, Hamad General Hospital., Doha, Baladīyat ad Dawḩah, Qatar

REFERENCES:
- [Background] Grissa MH, Claessens YE, Bouida W, Boubaker H, Boudhib L, Kerkeni W, Boukef R, Nouira S. Paracetamol vs piroxicam to relieve pain in renal colic. Results of a randomized controlled trial. Am J Emerg Med. 2011 Feb;29(2):203-6. doi: 10.1016/j.ajem.2009.09.019. Epub 2010 Oct 8. PMID 20934829
- [Background] Behzadnia MJ, Javadzadeh HR, Saboori F. Time of admission, gender and age: challenging factors in emergency renal colic - a preliminary study. Trauma Mon. 2012 Fall;17(3):329-32. doi: 10.5812/traumamon.6800. Epub 2012 Oct 10. PMID 24350118
- [Background] Shaden Salameh; Nurit Hiller; Meir Antopolsky; Fedaa Ghanem; Yigaal Abramovitz; Ruth Stalnikowics. Diclofenac versus Tramadol in the Treatment of Renal Colic: A Prospective, Randomized Trial. The Open Emergency Medicine Journal. 2011; 4: 9-13.
- [Derived] Pathan SA, Mitra B, Straney LD, Afzal MS, Anjum S, Shukla D, Morley K, Al Hilli SA, Al Rumaihi K, Thomas SH, Cameron PA. Delivering safe and effective analgesia for management of renal colic in the emergency department: a double-blind, multigroup, randomised controlled trial. Lancet. 2016 May 14;387(10032):1999-2007. doi: 10.1016/S0140-6736(16)00652-8. Epub 2016 Mar 16. PMID 26993881